CLINICAL TRIAL: NCT05940480
Title: TCM Daoyin Therapy in Early Chronic Obstructive Pulmonary Disease: A Pilot Study
Brief Title: TCM Daoyin Therapy in Individuals At-risk for COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Changzheng Community Health Service Center of Putuo District, Shanghai (Unknown)
Responsible Party: Principal Investigator, Lu Ying, MM, assistant researcher, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZY(2021-2023)- 0105-08
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Diseases, Obstructive
Keywords: TCM Daoyin; at-risk for COPD; early COPD; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: This study is a 16-week, randomized controlled trial. Individuals at-risk for COPD are randomized to either TCM Daoyin intervention group or health education control group.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors were blinded to the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM Daoyin intervention group (Experimental): Participants randomized to TCM Daoyin intervention group receive health education plus a TCM Daoyin training program. The TCM Daoyin training program was a 16-week, instructor-led group training program.
  Interventions: Behavioral: TCM Daoyin; Behavioral: Health education
- Health education control group (Active Comparator): Participants randomized to the health education control group only receive health education and no additional training program.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: TCM Daoyin — The TCM Daoyin training program consisted of two 90-min training classes and at least five 30-min at-home practice sessions per week for 16-weeks. All sessions included 10 min of warmup and 10 min of cooldown.
  Other Names: Qigong
  Arms: TCM Daoyin intervention group
Behavioral: Health education — Health education is provided by doctor and nurse, including work, rest, diet and other basic programs.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common, preventable and treatable disease. The aim of prospective randomized study is to evaluate the effects of TCM Daoyin training on Individuals at-risk for COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide. Early prevention and treatment of COPD is crucial, but there is a lack of specific interventions for individuals at-risk for COPD in clinical guidelines. The study focuses on individuals at-risk for COPD (COPD-SQ≥16, current lung function failed to meet diagnostic criteria for COPD but with manifestations of early airflow limitation).

This is a two-group prospective, randomized, assessor-blinded trial, planning to enroll 60 participants (30 for TCM Daoyin intervention group receiving health education plus a TCM Daoyin training program, and 30 for health education control group only receiving health education).

TCM Daoyin is a form of mind-body exercise with a profound philosophical foundation rooted in Chinese culture. Previous researches have provided some evidence of beneficial effects on TCM Daoyin for COPD patients with an established diagnosis, such as Liuzijue and Baduanjin. However, the evidences of TCM Daoyin on patients with early COPD is limited. The aim of prospective randomized study is to evaluate the effects of TCM Daoyin training on individuals at-risk of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Subject at-risk for COPD (Chronic obstructive pulmonary disease screening questionnaire (COPD-SQ) score≥16; and pre-bronchodilator FEV1/FVC ≥ 0.70, or pre-bronchodilator FEV1/FVC<0.70 but post-bronchodilator FEV1/FVC ≥ 0.70).
* Aged 40 to 75, male or female.
* Subject has a clear mind and the ability to lead an independent life.
* Subject agrees to perform a blood-test.
* Subject agrees to participate in this study and sign to the informed consent.

Exclusion Criteria:

* Subject with acute exacerbation of COPD.
* Subject with respiratory infectious disease (e.g., tuberculosis, influenza, etc.) within 1 month.
* Subject with serious current unstable physical illness and mental illness.
* Subject with definite clinical diagnosis of Alzheimer's disease, or severe cognitive impairment.
* Subject is pregnant or lactating women.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung function | Change from Baseline lung function at 16 weeks
  Participants' lung function (FVC、FVC%、FEV1、FEV1%、FEV1/FVC) will be tested to identify air flow condition in both group.

SECONDARY OUTCOMES:
6-min walk distance(6MWD) | Change from Baseline 6MWD at 16 weeks
  The 6MWD is a well-established field exercise test to assess the functional exercise capacity in COPD clinical trials.
Immune function | Change from Baseline immune function at 16 weeks
  Venous blood will be collect to detect immunity function (IL-6, IL-8, IL-10 and biomarkers).
Depression, Anxiety and Stress Scale-21 item (DASS-21) | Change from Baseline DASS-21 at 16 weeks
  Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
St. George's Respiratory Questionnaire (SGRQ) | Change from Baseline SGRQ at 16 weeks
  Quality of Life will be assessed by St. George's Respiratory Questionnaire (SGRQ). The SGRQ is a disease-specific measure of health status for use in COPD. It has a 0 - 100 score; 0 as low symptoms (feeling better) and 100 as high symptoms (feeling worse). A 4-unit change is the minimum clinically important difference.
Adverse effects | 8 weeks
  During the intervention period, the doctors will ask specifically about, and record any adverse effect of the treatment that may have occurred.
Adverse effects | 16 weeks
  During the intervention period, the doctors will ask specifically about, and record any adverse effect of the treatment that may have occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoting Zhao, Study Chair — Shanghai Qigong Research Institute; Jie Li, Doctor, Study Director — Shanghai University of Traditional Chinese Medicine; Ying Lu, Master, Principal Investigator — Shanghai Qigong Research Institute
Locations (2):
- China (2):
  - Shanghai Qigong Research Institute, Shanghai, Shanghai Municipality
  - Changzheng Community Health Service Center of Putuo District, Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No